CLINICAL TRIAL: NCT02185638
Title: Appetite Suppression Effects of an Herbal Combination of Yerba maté, Guarana, Damiana (YGD), and 12 Other Herbal Components, Versus YGD Supplementation Alone
Acronym: YGD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Arne Astrup, Professor, Dr Med, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: B258
Record Dates: First submitted 2012-06-19; First posted 2014-07-09 (Estimated); Last update posted 2014-07-09 (Estimated); Status verified 2014-07

CONDITIONS: Obesity
Keywords: obesity; herbal bioactive compounds; appetite; GLP-1; ghrelin; CCK
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A20-50 (Experimental): A20-50 (2 capsules). Each capsule contains:
  Yerba Mate (Ilex paraguariensis), Guarana seed (Paullinia cupana), Magnesium Oxide , Caffeine , Damiana (Turnera microphylla), Green tea (Camellia sinensis), Ginger (Zingiber Officinale), Kola nut (Cola acuminate or nitida), Pyridoxine Hydrochloride, Tibetan Ginseng root (Rhodiola crenulata), Schisandra (Schisandra Chinensis), Jujube (Ziziphus Jujuba) , Cocoa nut (Theobroma cacao), Chinese Skullcap (Scutellaria Baicalensis), Black tea leaf (Thea sinensis), Rice flour (to fill)
  Dose = 2 capsules have a total of 200 mg of caffeine
  Interventions: Other: Appetite suppressant properties of YGD and A20-50
- YGD (Active Comparator): YGD blend (2 capsules). Each capsule contains:
  Yerba Maté (leaf) , Guarana (seed) , Damiana (leaf) , Rice flour: to fill ,
  The 2 capsules of the YGD blend contain about 40 mg xanthines (caffeine and caffeine-like stimulants).
  Interventions: Other: Appetite suppressant properties of YGD and A20-50
- Placebo (Placebo Comparator): Placebo (2 capsules). Each capsule contains:
  Rice Flour
  Interventions: Other: Appetite suppressant properties of YGD and A20-50

INTERVENTIONS:
Other: Appetite suppressant properties of YGD and A20-50 — 3-arm crossover study for investigation of the effect of herbal supplements A20-50 compared to YGD blend and placebo on subjective appetite sensations, glucose, insulin, ghrelin, GLP-1, CCK and ad libitum energy intake

SUMMARY:
Background:

Supplementation with the combination of Yerba maté, guarana and damiana (YGD) has been found to slow gastric emptying by 15 to 58%, and to induce a substantial weight loss over 45 days without changes in diet. Enhanced gastric emptying rate has been shown to reduce the satiating effect of food and may thereby promote obesity. Yerba maté and guarana are known to contain large amounts of caffeine, resins, saponins and tannins, whereas damiana contains ethereal oils, tannins and resins. Caffeine belongs to a class of compounds called methylxanthines and epidemiological studies suggest that caffeine might possess weight reducing properties. The sympathomimetic properties of caffeine act to some extent through α- and β-adrenoreceptors, but most of the sympathoadrenergic stimulation caused by caffeine (even in very small doses) acts through the dual ability to antagonise adenosine and to inhibit the activity of cellular cyclic nucleotide phosphodiesterase. Stimulation of the sympathetic nervous system can cause suppression of hunger, enhance satiety and increase of energy expenditure covered in part by increased fat oxidation.

Aim:

To evaluate the effect of YGD combination or Akavar 20-50 (A20-50) compared with placebo on:

1. Acute change in 4-h subjective appetite sensations
2. Acute change in ad libitum energy intake (EI) 30 minutes post intake
3. Acute change in serum glucose, insulin, ghrelin and other appetite-regulating hormones (glucagon-like peptide-1 (GLP-1), cholecystokinin (CCK))

Subjects:

19 , healthy, premenopausal, overweight to obese (BMI between 27 and 32 kg/m2) women(age: 18 to 45 years).

Method:

The study is designed as a 3-way crossover, randomized, placebo controlled, double-blind study.

The bioactive components will be administered as capsules containing YGD or A20-50. The placebo capsules will contain rice flower. The subjects will undergo following treatments:

1. YGD capsules
2. A20-50 capsules
3. Placebo capsules

On each test day the subjects will be instructed to rest in a supine position for 15 minutes before dual measures of blood pressure and HR. A blood sample will be taken (baseline). The subject's appetite sensations will also be assessed by visual analogue scales (VAS) prior to intake of the test compound. Immediately hereafter the subjects will be served the first dose of the test compound. Blood samples will be taken at 15 and 30 minutes (time 0) post test compound. After 30 minutes post test compound the subjects will be given a standard breakfast (2.5 MJ = 598 kcal). Additional blood samples will be taken 15 minutes 30, 45, 60, 90, 120, 150, 180 and 240 minutes post-meal, together with a VAS appetite score assessment (0, 30, 45, 60, 90, 120, 150, 180 and 240 minutes).

Immediately after the last blood collection subjects will be asked to take a second dose of the test compound. After 30 minutes the subjects will repeat one VAS score assessment and be served an ad libitum lunch.

Blood samples will be analyzed for insulin, glucose, and appetite regulating hormones such as glucagon-like peptide-1 (GLP-1), ghrelin, cholecystokinin (CCK).

ELIGIBILITY:
Inclusion Criteria:

* Healthy,
* BMI: 27-32 kg/m2,
* Weight stable (within +/- 3 kg) two months prior to study inclusion,
* Non-smoking,
* Nonathletic (< 10 h hard physical activity),

Exclusion Criteria:

* BMI <27 and > 32 kg/m2,
* Change in smoking status,
* Daily or frequent use of medication,
* Suffering from metabolic diseases,
* Suffering from psychiatric diseases,
* Suffering from any other clinical condition, which would make the subject unfit to participate in the study,
* Hemoglobin < 7.0 mmol/l.
* alcohol and drug abuse
* blood donation, 3mo prior to the present study and during study participation

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Acute 3-h changes from baseline in subjective appetite sensations using visual analogue scales | Measured on 3 seperate test days in a crossover design. Each test day is seperated by >4 weeks. On each test day appetite sensations are measured prior to the test compound (time 0) and 30, 45, 60, 90, 120, 150, 180 and 240 minutes post intake
  Assessment of subjective appetite sensations (visual analogue scales (VAS)) at time 0 (baseline - prior to the test meal) and at time 30, 45, 60, 90, 120, 150, 180 and 240 minutes post intake.
  Measured subjective appetite sensations of hunger, satiety, prospective consumption, fullness, composite appetite score.

SECONDARY OUTCOMES:
Acute 3-h changes from baseline in subjective sensory desires using visual analogue scales | Measured on 3 seperate test days in a crossover design. Each test day is seperated by >4 weeks. On each test day appetite sensations are measured prior to the test compound (time 0) and 30, 45, 60, 90, 120, 150, 180 and 240 minutes post intake
  Assessment of subjective appetite sensations (visual analogue scales (VAS)) at time 0 (baseline - prior to the test meal) and at time 30, 45, 60, 90, 120, 150, 180 and 240 minutes post intake.
  Measured subjective sensory desires for something sweet, salty, rich in fat, or meat/fish
Acute 3-h changes from baseline in the postprandial concentration of Ghrelin | Measured on 3 seperate test days. Each test day is seperated by >4 weeks. Ghrelin was measured prior to the test compound (time -15 and -30 min) and to the breakfast meal (time 0) and 30, 45, 60, 90, 120, 150, 180 and 240 minutes
  A venflon catheter was secured into the participants' antecubital vein, and a blood sample was taken (baseline). Immediately after the subjects were served the test compound (2 capsules). Blood samples were taken at 15 and 30 minutes after intake of the test compound (2 capsules). After 30 minutes post test compound consumption (time 0), the subjects were given a standard breakfast (2.0 MJ: bun with cheese, yoghurt, 200 ml orange juice). Additional blood samples were taken 15, 30, 45, 60, 90, 120, 150, 180 and 240 minutes post-meal
Acute 3-h changes from baseline in the postprandial concentration of GLP-1 | Measured on 3 seperate test days. Each test day is seperated by >4 weeks. GLP-1 was measured prior to the test compound (time -15 and -30 min) and to the breakfast meal (time 0) and 30, 45, 60, 90, 120, 150, 180 and 240 minutes
  A venflon catheter was secured into the participants' antecubital vein, and a blood sample was taken (baseline). Immediately after the subjects were served the test compound (2 capsules). Blood samples were taken at 15 and 30 minutes after intake of the test compound (2 capsules). After 30 minutes post test compound consumption (time 0), the subjects were given a standard breakfast (2.0 MJ: bun with cheese, yoghurt, 200 ml orange juice). Additional blood samples were taken 15, 30, 45, 60, 90, 120, 150, 180 and 240 minutes post-meal
Acute 3-h changes from baseline in the postprandial concentration of CCK | Measured on 3 seperate test days. Each test day is seperated by >4 weeks. CCK was measured prior to the test compound (time -15 and -30 min) and to the breakfast meal (time 0) and 30, 45, 60, 90, 120, 150, 180 and 240 minutes
  A venflon catheter was secured into the participants' antecubital vein, and a blood sample was taken (baseline). Immediately after the subjects were served the test compound (2 capsules). Blood samples were taken at 15 and 30 minutes after intake of the test compound (2 capsules). After 30 minutes post test compound consumption (time 0), the subjects were given a standard breakfast (2.0 MJ: bun with cheese, yoghurt, 200 ml orange juice). Additional blood samples were taken 15, 30, 45, 60, 90, 120, 150, 180 and 240 minutes post-meal
Acute 3-h changes from baseline in the postprandial concentration of glucose | Measured on 3 seperate test days. Each test day is seperated by >4 weeks. Glucose was measured prior to the test compound (time -15 and -30 min) and to the breakfast meal (time 0) and 30, 45, 60, 90, 120, 150, 180 and 240 minutes
  A venflon catheter was secured into the participants' antecubital vein, and a blood sample was taken (baseline). Immediately after the subjects were served the test compound (2 capsules). Blood samples were taken at 15 and 30 minutes after intake of the test compound (2 capsules). After 30 minutes post test compound consumption (time 0), the subjects were given a standard breakfast (2.0 MJ: bun with cheese, yoghurt, 200 ml orange juice). Additional blood samples were taken 15, 30, 45, 60, 90, 120, 150, 180 and 240 minutes post-meal
Acute 3-h changes from baseline in the postprandial concentration of insulin | Measured on 3 seperate test days. Each test day is seperated by >4 weeks. Insulin was measured prior to the test compound (time -15 and -30 min) and to the breakfast meal (time 0) and 30, 45, 60, 90, 120, 150, 180 and 240 minutes
  A venflon catheter was secured into the participants' antecubital vein, and a blood sample was taken (baseline). Immediately after the subjects were served the test compound (2 capsules). Blood samples were taken at 15 and 30 minutes after intake of the test compound (2 capsules). After 30 minutes post test compound consumption (time 0), the subjects were given a standard breakfast (2.0 MJ: bun with cheese, yoghurt, 200 ml orange juice). Additional blood samples were taken 15, 30, 45, 60, 90, 120, 150, 180 and 240 minutes post-meal
Change in ad libitum energy intake (EI) | Measured on 3 seperate test days. Each test day is seperated by >4 weeks. EI was measured 240 min after intake of the breakfast meal.
  240 min after each test meal an ad libitum meal was served, and the total energy intake was recorded
Rating of the organoleptic quality of the ad libitum meal | Measured on 3 seperate test days. Each test day is seperated by >4 weeks.On each test day after completion of the ad libitum meal (approximately) time 15-20 minutes post intake) subjects will rate the ad libitum meal
  After completion of the adlibitum meal the subjects will rate the organoleptic quality of the meal by visual analogue scales (VAS) in regard to appearance, smell, taste, after-taste, and general palatability.
Subjective appetite sensations (visual analogue scales) after ad libitum meal | Measured on 3 seperate test days. Each test day is seperated by >4 weeks.After completion of the ad libitum meal subjects will rate their subjective sensation of appetite
  After completion of the ad libitum meal the subjects will rate the subjective appetite sensations by visual analogue scales (VAS) in regard to sensation of hunger, satiety, prospective consumption, fullness, composite appetite score and sensory desires to eat something sweet, salty, rich in fat, or meat/fish.
change in body weight | Measured on 3 seperate test days. Each test day is seperated by >4 weeks.On each test day body weight is carried out prior to the test.
  body weight will be measured to the nearest 0.05 kg on a decimal scale.
change in heart rate | Measured on 3 seperate test days. Each test day is seperated by >4 weeks.On each test day blood pressure and heart rate carried out prior to the test.
  heart rate were measured using an automatically inflating cuff.
change in blood pressure | Measured on 3 seperate test days. Each test day is seperated by >4 weeks.On each test day blood psure and heart rate carried out prior to the test.
  blood pressure were measured using an automatically inflating cuff.
change in composition (fat mass and fat free mass) | Measured on 3 seperate test days. Each test day is seperated by >4 weeks.On each test day composition is carried out prior to the test.
  Body composition will be assessed by electric bioimpedance using an Animeter.

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Professor, Dr Med, Principal Investigator — Department of Human Nutrition, Faculty of Science, University of Copenhagen, Denmark
Locations (1):
- Department Of Human Nutrition, Faculty of Science, University of Copenhagen, Frederiksberg, Denmark